CLINICAL TRIAL: NCT03966664
Title: Determination of Ka of Isolated Plasma and Whole Blood of Critically Ill Patients With Sepsis, Non-septic Patients and Healthy Volunteers: an International, In-vitro Acid-base Study.
Brief Title: Determination of the Dissociation Constant (Ka) of Plasma and Whole Blood in Septic Patients
Acronym: ENTERPRISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: ENTERPRISE
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Sepsis; Septic Shock; Critical Illness; Respiratory Acidosis; Respiratory Alkalosis; Acid-Base Imbalance
Keywords: Acid-base equilibrium; pH; septic shock; critical illness
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness; Acidosis, Respiratory; Alkalosis, Respiratory; Acid-Base Imbalance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples in ethylenediaminetetraacetic acid for subsequent biomolecular analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Septic patients: Critically ill patients of both sexes admitted to the general ICU of the participating centers with the diagnosis of sepsis will be included.
  Interventions: Diagnostic Test: In vitro determination the dissociation constant (Ka) and total amount of non-volatile buffers (Atot) in isolated plasma.; Diagnostic Test: In vitro determination the dissociation constant (Ka) and total amount of non-volatile buffers (Atot) in whole blood; Diagnostic Test: Biomolecular analysis of plasma proteins.
- Healthy controls: Age and sex matched healthy volunteers.
  Interventions: Diagnostic Test: In vitro determination the dissociation constant (Ka) and total amount of non-volatile buffers (Atot) in isolated plasma.; Diagnostic Test: In vitro determination the dissociation constant (Ka) and total amount of non-volatile buffers (Atot) in whole blood; Diagnostic Test: Biomolecular analysis of plasma proteins.
- Non septic patients: Non-septic patients admitted to the general ICU of the participating centers after elective non-cardiac surgery.
  Interventions: Diagnostic Test: In vitro determination the dissociation constant (Ka) and total amount of non-volatile buffers (Atot) in isolated plasma.; Diagnostic Test: In vitro determination the dissociation constant (Ka) and total amount of non-volatile buffers (Atot) in whole blood; Diagnostic Test: Biomolecular analysis of plasma proteins.

INTERVENTIONS:
Diagnostic Test: In vitro determination the dissociation constant (Ka) and total amount of non-volatile buffers (Atot) in isolated plasma. — Collection of a venous blood sample, centrifugation in order to harvest isolated plasma and performance of in-vitro tonometry in order to assess Ka and Atot.
Diagnostic Test: In vitro determination the dissociation constant (Ka) and total amount of non-volatile buffers (Atot) in whole blood — Collection of a venous blood sample and performance of in-vitro tonometry in order to assess Ka and Atot.
Diagnostic Test: Biomolecular analysis of plasma proteins. — Bidimensional electrophoresis, determination of oxidized albumin fraction, characterization of altered ligand binding properties of plasma albumin.

SUMMARY:
Alterations of acid-base equilibrium are very common in critically ill patients and understanding their pathophysiology can be important to improve clinical treatment.

DETAILED DESCRIPTION:
Acid-base equilibrium has been object of study for more than 100 years in medicine because of its relevance in patients' management and in determining their prognosis, especially in the ICU.

A concept closely related to acid-base equilibrium is that of "buffer", term used to define any substance able to limit the changes in pH caused by the addition or loss of alkali or acid.

Depending on its physiochemical features, every buffer has one or more pH (negative logarithm of hydrogen ion concentration) values where its ability to keep pH stable is maximal. These values are defined as Ka or semi equivalence points, i.e. the pH values where the buffer dissolved in solution is half in its associated form (AH) and half in its dissociated form (A-).

Several studies tried to determine the normal values of both concentration and Ka of ATOT. However, they did not lead to univocal results. Moreover, many of these values come from studies of veterinary medicine or are the result of theoretical estimates on human plasma.

Staempfli and Constable performed a single experimental study on human plasma in 2003. These authors, however, analyzed only isolated plasma, neglecting whole blood, and computed ATOT and Ka values of healthy volunteers, while Ka and ATOT values for critically ill patients with sepsis are still unknown.

Primary aim of the present study is to quantify the acidic dissociation constant (Ka) of isolated plasma of critically ill patients with sepsis, and compare these data with normal values, i.e. obtained from healthy controls. The investigators hypothesize that plasma of critically ill septic patients has a lower Ka and that, consequently, it undergoes higher pH variations for a given perturbation of the system (variation in carbon dioxide).

Secondary aim is to quantify the Ka of whole blood of critically ill patients with sepsis and compare these data with normal values, i.e. obtained from healthy controls. The investigators hypothesize that blood of critically ill septic patients has a lower Ka and that, consequently, it undergoes higher pH variations for a given perturbation of the system (variation in carbon dioxide).

Other aims of the study are:

* quantify the Ka of plasma and whole blood of non-septic patients admitted to the ICU and compare these results with the values of septic patients and healthy volunteers.
* define the normal concentration of weak non-carbonic acids (ATOT) in plasma of septic patients and compare it with data obtained in healthy volunteers and non-septic patients.

Finally, possible structural alteration of plasma proteins will be evaluated:

* Identification of differentially modified proteoforms of serum albumin and major plasma proteins by two-dimensional electrophoresis;
* High Performance Liquid Chromatography (HPLC) to identify different Redox-forms of albumin
* Spectrophotometric evaluation of modifications of ligand binding properties of serum albumin.

ELIGIBILITY:
Group 1: Septic patients

Inclusion Criteria for Group 1:

* Diagnosis of Sepsis
* Age > 18 years
* Informed or deferred informed consent

Exclusion Criteria for Group 1:

* Pregnancy
* Bilirubin > 4 mg/dL
* Minor or major thalassemia
* Transfusion of more than 4 Units of packed red blood cells and/or 1 L of plasma during the 24 hours prior to enrollment

Group 2: Healthy volunteers

Inclusion criteria for Group 2:

* informed consent
* Age > 18 years

Exclusion criteria for Group 2:

• Pregnancy

Group 3: Non-septic patients

Inclusion criteria for Group 3:

* Informed consent
* Age >18 years
* Planned ICU admission after elective surgery

Exclusion criteria for Group 3:

* Diagnosis of sepsis
* Pregnancy
* Bilirubin >4 mg/dL
* Liver cirrhosis
* Onco-hematological diseases
* Minor or major thalassemia
* Transfusion of more than 4 Units of packed red blood cells and/or 1 L of plasma during the 24 hours prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with sepsis or septic shock admitted to the ICU
  2. Healthy volunteers recruited from ICU staff members and relatives
  3. Non-septic patients admitted to the ICU after elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Effective dissociation constant of plasma weak acids (Ka) [dimensionless] | 1 day
  Difference in plasma Ka between study groups.

SECONDARY OUTCOMES:
Effective dissociation constant of whole blood weak acids (Ka) [dimensionless] | 1 day
  Difference in whole blood Ka between study groups.
Total concentration of plasma non-volatile buffers (Atot) [mmol/L] | 1 day
  Difference in plasma Atot between study groups.
Total concentration of whole blood non-volatile buffers (Atot) [mmol/L] | 1 day
  Difference in whole blood Atot between study groups.
Non-carbonic buffer power of whole blood due to electrolyte shifts [milliequivalents/L] | 1 day
  Difference in Non-carbonic buffer power of whole blood due to electrolyte shifts between study groups.
Non-carbonic buffer power of isolated plasma due to electrolyte shifts [milliequivalents/L] | 1 day
  Difference in Non-carbonic buffer power of isolated plasma due to electrolyte shifts between study groups.
Oxidized albumin [%] | 1 day
  Difference in the percentage in oxidized albumin between groups.
Characterization of altered ligand binding properties | 1 day
  HSA will be fractionated and dissociation constants for warfarin-SA and diazepam-SA complexes will be obtained spectrophotometrically to evaluate modifications in its ligand binding properties
Identification of differentially modified proteoforms of human serum albumin (HSA) and major plasma proteins. | 1 day
  Samples will be analyzed by two-dimensional electrophoresis.8 After fluorescent staining and image acquisition, proteoform patterns corresponding to HSA and other major plasma proteins will be aligned and compared

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Langer, MD, Principal Investigator — Fondazione IRCCS Ca' Granda Hospital, Milano, Italy; Antonio M Pesenti, MD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Frantisek Duska, MD, Principal Investigator — Third faculty of Medicine, Charles University, Prague; Giacomo Grasselli, MD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Paul Elbers, MD, Study Chair — Amsterdam UMC, Department of Intensive Care Medicine
Locations (2):
- Third faculty of Medicine, Charles University of Prague, Prague, Czechia
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Background] Henderson LJ. THE REGULATION OF NEUTRALITY IN THE ANIMAL BODY. Science. 1913 Mar 14;37(950):389-95. doi: 10.1126/science.37.950.389. No abstract available. PMID 17795147
- [Background] Lee SW, Hong YS, Park DW, Choi SH, Moon SW, Park JS, Kim JY, Baek KJ. Lactic acidosis not hyperlactatemia as a predictor of in hospital mortality in septic emergency patients. Emerg Med J. 2008 Oct;25(10):659-65. doi: 10.1136/emj.2007.055558. PMID 18843064
- [Background] Fencl V, Leith DE. Stewart's quantitative acid-base chemistry: applications in biology and medicine. Respir Physiol. 1993 Jan;91(1):1-16. doi: 10.1016/0034-5687(93)90085-o. PMID 8441866
- [Background] LEEUWEN AM. NET CATION EQUIVALENCY ('BASE BINDING POWER') OF THE PLASMA PROTEINS. Acta Med Scand. 1964;176:SUPPL 422: 1+. No abstract available. PMID 14204741
- [Background] Figge J, Mydosh T, Fencl V. Serum proteins and acid-base equilibria: a follow-up. J Lab Clin Med. 1992 Nov;120(5):713-9. PMID 1431499
- [Background] Stampfli HR, Misiaszek S, Lumsden JH, Carlson GP, Heigenhauser GJ. Weak acid-concentration Atot and dissociation constant Ka of plasma proteins in racehorses. Equine Vet J Suppl. 1999 Jul;(30):438-42. PMID 10659296
- [Background] Staempfli HR, Constable PD. Experimental determination of net protein charge and A(tot) and K(a) of nonvolatile buffers in human plasma. J Appl Physiol (1985). 2003 Aug;95(2):620-30. doi: 10.1152/japplphysiol.00100.2003. Epub 2003 Mar 28. PMID 12665532
- [Background] Langer T, Scotti E, Carlesso E, Protti A, Zani L, Chierichetti M, Caironi P, Gattinoni L. Electrolyte shifts across the artificial lung in patients on extracorporeal membrane oxygenation: interdependence between partial pressure of carbon dioxide and strong ion difference. J Crit Care. 2015 Feb;30(1):2-6. doi: 10.1016/j.jcrc.2014.09.013. Epub 2014 Sep 22. PMID 25307980